CLINICAL TRIAL: NCT01473758
Title: Effect of Roflumilast 500 μg Tablets Once Daily at Acute COPD Exacerbations Treated With Standard Therapy of Oral Steroids and Antibiotics. A Randomised, Double-blind, Placebo-controlled, Parallel-group Trial
Brief Title: Effect of Roflumilast at Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Acronym: TREAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision: No Safety or Efficacy Concerns
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO-2455-405-RD; 2011-002905-31 (EudraCT Number); U1111-1137-4023 (Registry Identifier: WHO); 11/SC/0494 (Registry Identifier: NRES)
Record Dates: First submitted 2011-10-31; First posted 2011-11-17 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-08

CONDITIONS: Chronic Obstructive Pulmonary Disease With (Acute) Exacerbation
Keywords: COPD; Chronic obstructive pulmonary disease; Roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Active Comparator): added on to standard therapy for acute COPD exacerbations
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): added on to standard therapy for acute COPD exacerbations
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 µg tablet, od, oral administration in the morning after breakfast
  Arms: Roflumilast
Drug: Placebo — tablet, od, oral administration in the morning after breakfast
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate if roflumilast can reduce the neutrophilic inflammation at acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD). In addition, the potential benefit of roflumilast on severity and recovery periods of acute COPD exacerbations will be assessed using patient diaries and questionnaires.

DETAILED DESCRIPTION:
Participants will be asked whether they agree to participate in the measurements of arterial stiffness. Participants who agree will be included in the substudy, with the target of 60 patients with arterial stiffness measurements to complete the trial.

Study was terminated due to difficulty in identifying further eligible patients for this exploratory study within a reasonable time.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC)
* Age ≥ 40 years
* History of COPD for at least 12 months prior to enrollment (Visit V0)
* Chronic productive cough for 3 months in each of the 2 years prior to enrollment (if other causes of productive cough have been excluded) and/or an exacerbation with predominantly bronchitic symptoms at enrollment
* Presentation of an acute exacerbation of COPD that will be associated with increased sputum volume or change in sputum colour
* Documented fixed airway obstruction determined by an FEV1/FVC ratio (post-bronchodilator) < 70% (if a pulmonary function test is not possible at Visit V0 a previous measurement can be taken which must not be older than 6 months)
* Former smoker (defined as: smoking cessation at least 1 year ago) or current smoker both with a smoking history of at least 10 pack years

Main Exclusion Criteria:

* Diagnosis of asthma and/or other relevant lung disease
* Known alpha-1-antitrypsin deficiency
* Recurrent exacerbations (within 8 weeks of a preceding exacerbation)
* Treatment of current exacerbation with oral corticosteroids and/or antibiotics already started at enrollment
* Treatment with PDE4 inhibitors within 3 months prior to Visit V0
* Other protocol-defined exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- United Kingdom (2):
  - Academic Unit of Respiratory Medicine, Royal Free Hospital, Jadwiga A. Wedzicha, London
  - London

REFERENCES:
- [Derived] Mackay AJ, Patel ARC, Singh R, Sapsford RJ, Donaldson GC, Prasad N, Goehring UM, Nip TK, Wedzicha JA. Randomized Double-Blind Controlled Trial of Roflumilast at Acute Exacerbations of Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Sep 1;196(5):656-659. doi: 10.1164/rccm.201612-2518LE. No abstract available. PMID 28146642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 16 February 2012 to 25 March 2014.
Pre-assignment Details: Participants with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) were enrolled equally in 1 of 2 treatment groups, once a day placebo or roflumilast 500 µg in Cycle 1. Participants were re-randomized in Cycle 2 to once a day placebo or roflumilast 500 µg and are counted as new participants.
Groups:
- Roflumilast 500 μg: Roflumilast 500 µg tablet, once daily, orally in the morning after breakfast for 4 weeks added on to standard therapy for acute COPD exacerbations. Eligible participants were re-randomized to receive either roflumilast 500 μg or placebo for 4 weeks in Cycle 2.
- Placebo: Placebo matching roflumilast tablet, once daily, orally in the morning after breakfast added on to standard therapy for acute COPD exacerbations. Eligible participants were re-randomized to receive either roflumilast 500 μg or placebo for 4 weeks in Cycle 2.
- Roflumilast 500 µg (Cycle 2): Roflumilast 500 µg tablet, once daily, orally in the morning after breakfast for 4 weeks added on to standard therapy for acute COPD exacerbations in Cycle 2.
- Placebo (Cycle 2): Placebo matching roflumilast tablet, once daily, orally in the morning after breakfast for 4 weeks added on to standard therapy for acute COPD exacerbations in Cycle 2.
Period: Cycle 1
Arm/Group | Roflumilast 500 μg | Placebo | Roflumilast 500 µg (Cycle 2) | Placebo (Cycle 2)
Started | 38 | 43 | 0 | 0
Completed | 27 | 40 | 0 | 0
Not Completed | 11 | 3 | 0 | 0
Not completed — Adverse Event | 10 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Period: Cycle 2
Arm/Group | Roflumilast 500 μg | Placebo | Roflumilast 500 µg (Cycle 2) | Placebo (Cycle 2)
Started | 0 | 0 | 10 | 4
Completed | 0 | 0 | 5 | 4
Not Completed | 0 | 0 | 5 | 0
Not completed — Adverse Event | 0 | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis set consisted of all randomized patients who received at least 1 dose of investigational medicinal product (IMP)
Groups:
- Roflumilast 500 μg: Roflumilast 500 µg tablet, once daily, orally in the morning after breakfast for 4 weeks added on to standard therapy for acute COPD exacerbations.
- Placebo: Placebo matching roflumilast tablet, once daily, orally in the morning after breakfast for 4 weeks added on to standard therapy for acute COPD exacerbations.
- Total: Total of all reporting groups
Arm/Group | Roflumilast 500 μg | Placebo | Total
Number analyzed (Participants) | 38 | 43 | 81
Age, Customized [Number; unit: participants]
  ≤ 65 years | 7 | 11 | 18
  > 65 years | 31 | 32 | 63
Gender [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 22 | 28 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 1 | 3
  White | 36 | 42 | 78
Smoking status [Number; unit: participants]
  Non-smoker | 0 | 0 | 0
  Current smoker | 8 | 11 | 19
  Former smoker | 30 | 32 | 62
Baseline COPD Assessment Test (CAT) Total Score [Number; unit: participants] — The CAT is a short, validated, patient-completed questionnaire to assess the impact of COPD on health status. It comprises 8 questions that cover a broad range of effects of COPD on patients' health. Each question is scored in a range between 0 and 5, with the higher end indicating a higher impact of COPD on the patient's wellbeing. The CAT Total score ranges from 0 best) to 40 (Worst).
  participants
    < 10 | 2 | 3 | 5
    ≥ 10 | 16 | 25 | 41
    Missing | 20 | 15 | 35
Weight Category by Body Mass Index (BMI) [Number; unit: participants]
  Underweight | 3 | 0 | 3
  Normal Weight | 15 | 18 | 33
  Overweight | 11 | 15 | 26
  Obese | 9 | 9 | 18
  Missing | 0 | 1 | 1
Chronic Bronchitis [Number; unit: participants]
  No | 14 | 17 | 31
  Yes | 24 | 26 | 50
Historical Chronic Obstructive Pulmonary Disease (COPD) Exacerbations [Number; unit: participants]
  < 2 | 28 | 28 | 56
  ≥ 2 | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sputum Neutrophil Counts at Day 14 Post Exacerbation (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Total cell count (absolute number of nonsquamous cells per gram of the original sputum sample) were determined using a Neubauer hemocytometer. A negative change from Baseline indicates improvement. An Analysis of Covariance (ANCOVA) model was used with neutrophil count at Baseline and treatment as independent variables, fixed effects.
Time Frame: Baseline and Day 14
Population: Participants from the Intent-to-treat (ITT) population, all randomized participants, with data available at the given time-point. Analysis included all participants who received treatment in Cycle 1.
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/gram sputum
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 29 | 37
10^6 cells/gram sputum | -18.705 (2.263) | -20.109 (1.995)
Statistical Analysis 1: Comparison: Roflumilast 500 μg vs Placebo; Test type: Superiority or Other; p = 0.6491, ANCOVA — The model contains neutrophil count at Baseline and treatment as independent variables, fixed effects; LS Mean Difference = 1.404, 95% CI 2-sided [-4.731 to 7.538], Standard Error of Mean 3.070

2. Primary Outcome: Change From Baseline in Sputum Neutrophil Counts at Day 14 Post Exacerbation (Extended Approach)
Description: as for outcome 1
Time Frame: Baseline and Day 14
Population: Participants from the Intent-to-treat population, all randomized participants, with data available at the given time-point. Extended Approach Analysis included all participants who received treatment in Cycle 1 and participants who were re-randomized and received treatment in Cycle 2.
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/gram sputum
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 37 | 39
10^6 cells/gram sputum | -19.569 (1.906) | -19.157 (1.855)
Statistical Analysis 1: Comparison: Roflumilast 500 μg vs Placebo; Test type: Superiority or Other; p = 0.8786, ANCOVA — The model contains neutrophil count at Baseline and treatment as independent variables, fixed effects; LS Mean Difference = -0.412, 95% CI 2-sided [-5.766 to 4.943], Standard Error of Mean 2.687

3. Secondary Outcome: Percentage of Participants Whose Sputum Neutrophil Counts Returned to Stable State at Day 14 (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Total cell count (absolute number of nonsquamous cells per gram of the original sputum sample) and were determined with a Neubauer hemocytometer.
Time Frame: Day 14
Population: Participants from the Intent-to-treat (ITT) population, all randomized participants, with data available at the given time-point. Initial Approach Analysis included all participants who received treatment in Cycle 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 16 | 29
percentage of participants | 37.5 [15.2 to 64.6] | 55.2 [35.7 to 73.6]

4. Secondary Outcome: Percentage of Participants Whose Sputum Neutrophil Counts Returned to Stable State at Day 14 (Extended Approach)
Description: as for outcome 3
Time Frame: Day 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 20 | 31
percentage of participants | 45.0 [23.1 to 68.5] | 51.6 [33.1 to 69.8]

5. Secondary Outcome: Change From Baseline in Sputum Marker Total Cells (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Total cell count (absolute number of nonsquamous cells per gram of the original sputum sample) were determined using a Neubauer hemocytometer. A negative change from Baseline indicates improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/gram sputum
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
10^6 cells/gram sputum
  Change at Day 7 (n=35, 39) | -25.559 (3.529) | -27.563 (3.334)
  Change at Day 14 (n=32, 38) | -21.813 (2.706) | -25.111 (2.505)
  Change at Day 28 (n=25, 37) | -29.200 (4.022) | -22.218 (3.362)
  Change at Day 56 (n=24, 33) | -24.477 (2.708) | -26.474 (2.341)

6. Secondary Outcome: Change From Baseline in Sputum Marker Total Cells (Extended Approach)
Description: as for outcome 5
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/gram sputum
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 46
10^6 cells/gram sputum
  Change at Day 7 (n=45, 43) | -26.634 (3.030) | -26.335 (3.124)
  Change at Day 14 (n=41, 42) | -23.512 (2.448) | -25.332 (2.471)
  Change at Day 28 (n=30, 40) | -29.023 (3.347) | -22.920 (2.947)
  Change at Day 56 (n=28, 36) | -19.551 (3.920) | -26.855 (3.536)

7. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Neutrophils (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Aliquots of a cell suspension prepared from the sputum sample were used to prepare cytospin slides that were stained with Diff-Quik for differential cell counts. 100 cells were counted and the percentage of neutrophils was determined. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of neutrophils
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 43
percentage of neutrophils
  Change at Day 7 (n=30, 35) | -11.325 (3.837) | -14.484 (3.559)
  Change at Day 14 (n=31, 37) | -16.770 (3.983) | -20.346 (3.550)
  Change at Day 28 (n=24, 34) | -27.760 (5.275) | -13.837 (4.498)
  Change at Day 56 (n=16, 30) | -19.663 (5.561) | -17.047 (4.229)

8. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Neutrophils (Extended Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Aliquots of a cell suspension prepared from the sputum sample were used to prepare cytospin slides that were stained with Diff-Quik for differential cell counts. 100 cells were counted and the percentage of neutrophils was determined. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of neutrophils
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 46
percentage of neutrophils
  Change at Day 7 (n=37, 39) | -14.637 (3.748) | -16.060 (3.713)
  Change at Day 14 (n=39, 40) | -20.690 (3.758) | -21.052 (3.678)
  Change at Day 28 (n=29, 36) | -29.848 (4.721) | -14.664 (4.371)
  Change at Day 56 (n=20, 32) | -21.327 (5.009) | -17.328 (4.188)

9. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Macrophages (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Aliquots of a cell suspension prepared from the sputum sample were used to prepare cytospin slides that were stained with Diff-Quik for differential cell counts. 100 cells were counted and the percentage of macrophages was determined. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of macrophages
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 43
percentage of macrophages
  Change at Day 7 (n=30, 35) | 11.393 (3.837) | 15.430 (3.559)
  Change at Day 14 (n=31, 37) | 16.062 (3.929) | 20.774 (3.506)
  Change at Day 28 (n=24, 34) | 27.535 (5.284) | 13.382 (4.503)
  Change at Day 56 (n=16, 30) | 16.593 (5.539) | 15.877 (4.171)

10. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Macrophages (Extended Approach)
Description: as for outcome 9
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of macrophages
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 46
percentage of macrophages
  Change at Day 7 (n=37, 39) | 14.679 (3.740) | 17.228 (3.704)
  Change at Day 14 (n=39, 40) | 20.331 (3.745) | 21.599 (3.667)
  Change at Day 28 (n=29, 36) | 29.510 (4.717) | 14.463 (4.367)
  Change at Day 56 (n=20, 32) | 19.075 (5.003) | 16.322 (4.156)

11. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Eosinophils (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Aliquots of a cell suspension prepared from the sputum sample were used to prepare cytospin slides that were stained with Diff-Quik for differential cell counts. 100 cells were counted and the percentage of eosinophils was determined. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of eosinophils
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 43
percentage of eosinophils
  Change at Day 7 (n=30, 35) | -0.259 (0.245) | -0.100 (0.225)
  Change at Day 14 (n=31, 37) | -0.110 (0.326) | -0.188 (0.288)
  Change at Day 28 (n=24, 34) | 0.043 (1.209) | 1.597 (1.020)
  Change at Day 56 (n=16, 30) | 2.187 (2.278) | 1.086 (1.766)

12. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Eosinophils (Extended Approach)
Description: as for outcome 11
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of macrophages
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 46
percentage of macrophages
  Change at Day 7 (n=37, 39) | -0.341 (0.206) | -0.141 (0.202)
  Change at Day 14 (n=39, 40) | -0.174 (0.271) | -0.214 (0.263)
  Change at Day 28 (n=29, 36) | 0.031 (1.044) | 1.518 (0.952)
  Change at Day 56 (n=20, 32) | 1.714 (1.969) | 0.913 (1.655)

13. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Lymphocyte (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Aliquots of a cell suspension prepared from the sputum sample were used to prepare cytospin slides that were stained with Diff-Quik for differential cell counts. 100 cells were counted and the percentage of lymphocytes was determined. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of lymphocytes
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 43
percentage of lymphocytes
  Change at Day 7 (n=30, 35) | 0.229 (0.353) | 0.182 (0.326)
  Change at Day 14 (n=31, 37) | 0.430 (0.254) | 0.295 (0.225)
  Change at Day 28 (n=24, 34) | 0.039 (0.183) | -0.325 (0.155)
  Change at Day 56 (n=16, 30) | -0.095 (0.187) | -0.051 (0.137)

14. Secondary Outcome: Change From Baseline in Sputum Marker Percentage of Lymphocytes (Extended Approach)
Description: as for outcome 13
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of lymphocytes
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 46
percentage of lymphocytes
  Change at Day 7 (n=37, 39) | 0.109 (0.308) | -0.015 (0.303)
  Change at Day 14 (n=39, 40) | 0.309 (0.250) | 0.195 (0.243)
  Change at Day 28 (n=29, 36) | -0.118 (0.173) | -0.431 (0.158)
  Change at Day 56 (n=20, 32) | -0.203 (0.164) | -0.208 (0.132)

15. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Interleukin (IL)-6 (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Sputum inflammatory marker IL-6 was quantified by commercial sandwich enzyme-linked immunosorbent assays (ELISA). A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 42
pg/mL
  Change at Day 7 (n=31, 38) | -1317.400 (143.748) | -934.624 (133.217)
  Change at Day 14 (n=30, 35) | -822.715 (221.328) | -695.955 (206.201)
  Change at Day 28 (n=22, 35) | -1232.929 (212.663) | -955.365 (174.734)
  Change at Day 56 (n=22, 29) | -1042.097 (225.619) | -996.485 (196.729)

16. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Interleukin (IL)-6 (Extended Approach)
Description: as for outcome 15
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 45
pg/mL
  Change at Day 7 (n=37, 42) | -1207.678 (133.298) | -923.325 (130.533)
  Change at Day 14 (n=36, 39) | -725.454 (195.921) | -705.849 (192.890)
  Change at Day 28 (n=26, 38) | -1115.741 (200.367) | -877.871 (172.950)
  Change at Day 56 (n=26, 32) | -860.191 (206.289) | -962.342 (189.817)

17. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Interleukin (IL)-8 (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Sputum inflammatory marker IL-8 was quantified by commercial sandwich enzyme-linked immunosorbent assays (ELISA). A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 42
pg/mL
  Change at Day 7 (n=31, 38) | -174718.396 (45481.710) | -227274.816 (41821.023)
  Change at Day 14 (n=30, 35) | -149198.139 (47388.834) | -199515.687 (43965.789)
  Change at Day 28 (n=22, 35) | -255317.294 (70915.154) | -160587.365 (57944.793)
  Change at Day 56 (n=21, 29) | -204731.356 (50404.332) | -223918.341 (43039.568)

18. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Interleukin (IL)-8 (Extended Approach)
Description: as for outcome 17
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 45
pg/mL
  Change at Day 7 (n=37, 42) | -193222.856 (39595.196) | -215296.477 (38432.424)
  Change at Day 14 (n=36, 39) | -172069.810 (41341.330) | -195751.307 (40449.866)
  Change at Day 28 (n=26, 38) | -264788.038 (62440.420) | -160441.028 (53963.528)
  Change at Day 56 (n=25, 32) | -168204.970 (51760.361) | -205822.814 (46476.985)

19. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Myeloperoxidase (MPO) (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Sputum inflammatory marker MPO was quantified by commercial sandwich enzyme-linked immunosorbent assays (ELISA). A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 42
ng/mL
  Change at Day 7 (n=31, 38) | -9253.786 (1997.077) | -4521.397 (1863.867)
  Change at Day 14 (n=30, 35) | -8072.784 (2144.895) | -6318.878 (2002.939)
  Change at Day 28 (n=22, 35) | -13744.824 (2476.123) | -5944.184 (2041.587)
  Change at Day 56 (n=22, 29) | -10248.612 (2578.146) | -9478.460 (2234.238)

20. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Myeloperoxidase (MPO) (Extended Approach)
Description: as for outcome 19
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 45
ng/mL
  Change at Day 7 (n=37, 42) | -8606.357 (1747.094) | -4380.803 (1713.047)
  Change at Day 14 (n=36, 39) | -8380.855 (1871.930) | -5929.775 (1843.806)
  Change at Day 28 (n=26, 38) | -12692.279 (2220.374) | -5351.001 (1933.964)
  Change at Day 56 (n=26, 32) | -9424.227 (2275.981) | -8527.766 (2078.411)

21. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Neutrophil Elastase (Initial Approach)
Description: Sputum samples were collected and processed at the investigational site according to their standard procedures. Sputum inflammatory marker Neutrophil Elastase was quantified by commercial sandwich enzyme-linked immunosorbent assays (ELISA). A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: µg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 36 | 42
µg/mL
  Change at Day 7 (n=31, 38) | -222995.020 (14887.254) | -224606.396 (13669.986)
  Change at Day 14 (n=30, 35) | -149211.318 (39523.470) | -125385.276 (36629.962)
  Change at Day 28 (n=22, 35) | -200905.068 (25432.984) | -149865.936 (20549.567)
  Change at Day 56 (n=21, 30) | -141985.838 (28278.566) | -169389.587 (23767.879)

22. Secondary Outcome: Change From Baseline in Sputum Marker Concentration of Neutrophil Elastase (Extended Approach)
Description: as for outcome 21
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: µg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 46 | 45
µg/mL
  Change at Day 7 (n=37, 42) | -202235.344 (12993.506) | -206912.465 (12543.143)
  Change at Day 14 (n=36, 39) | -143831.510 (34043.871) | -110144.325 (33211.578)
  Change at Day 28 (n=26, 38) | -183452.324 (22560.241) | -130613.019 (19255.852)
  Change at Day 56 (n=25, 33) | -118129.436 (25397.042) | -156544.533 (22550.054)

23. Secondary Outcome: Change From Baseline in Blood Biomarker Interleukin (IL)-6 (Initial Approach)
Description: Blood was collected and serum biomarker IL-6 was quantified using commercial sandwich ELISA. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
pg/mL
  Change at Day 7 (n=37, 41) | -12.469 (0.782) | -11.904 (0.742)
  Change at Day 14 (n=33, 41) | -1.973 (1.918) | -5.728 (1.730)
  Change at Day 28 (n=28, 40) | -8.108 (2.360) | -7.243 (1.997)
  Change at Day 56 (n=27, 40) | -11.665 (1.129) | -9.431 (0.937)

24. Secondary Outcome: Change From Baseline in Blood Biomarker Interleukin (IL)-6 (Extended Approach)
Description: as for outcome 23
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
pg/mL
  Change at Day 7 (n=47, 45) | -12.314 (0.652) | -11.802 (0.665)
  Change at Day 14 (n=43, 45) | 1.607 (2.543) | -6.069 (2.490)
  Change at Day 28 (n=33, 44) | -7.587 (2.088) | -7.619 (1.838)
  Change at Day 56 (n=32, 44) | -10.811 (1.064) | -9.604 (0.918)

25. Secondary Outcome: Change From Baseline in Blood Biomarker Interleukin-1 Beta (IL-1β) (Initial Approach)
Description: Blood was collected and serum biomarker IL-1β was quantified using commercial sandwich ELISA. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
pg/mL
  Change at Day 7 (n=37, 41) | 1.274 (0.682) | 0.378 (0.647)
  Change at Day 14 (n=33, 41) | 0.217 (0.359) | 0.495 (0.324)
  Change at Day 28 (n=28, 40) | 0.657 (0.431) | 0.541 (0.366)
  Change at Day 56 (n=27, 40) | -0.003 (0.329) | 0.464 (0.288)

26. Secondary Outcome: Change From Baseline in Blood Biomarker IL-1β (Extended Approach)
Description: as for outcome 25
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
pg/mL
  Change at Day 7 (n=47, 45) | 0.350 (0.590) | -1.002 (0.602)
  Change at Day 14 (n=43, 45) | -0.394 (0.355) | -0.841 (0.349)
  Change at Day 28 (n=33, 44) | -0.139 (0.414) | -0.757 (0.368)
  Change at Day 56 (n=32, 44) | -0.799 (0.333) | -0.806 (0.312)

27. Secondary Outcome: Change From Baseline in Blood Biomarker C-reactive Protein (CRP) (Initial Approach)
Description: Blood was collected and serum biomarker CRP was measured using Roche Modular Analytics E 170 Module. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/liter(L)
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
mg/liter(L)
  Change at Day 7 (n=37, 41) | -15.579 (0.485) | -16.518 (0.461)
  Change at Day 14 (n=33, 41) | 4.836 (4.249) | -4.369 (3.812)
  Change at Day 28 (n=28, 38) | -9.179 (4.110) | -8.018 (3.533)
  Change at Day 56 (n=26, 40) | -14.889 (1.395) | -13.057 (1.133)

28. Secondary Outcome: Change From Baseline in Blood Biomarker C-reactive Protein (CRP) (Extended Approach)
Description: as for outcome 27
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
mg/L
  Change at Day 7 (n=47, 45) | -16.166 (0.410) | -16.901 (0.417)
  Change at Day 14 (n=43, 45) | 5.720 (3.600) | -5.257 (3.518)
  Change at Day 28 (n=33, 42) | -8.250 (3.802) | -9.254 (3.375)
  Change at Day 56 (n=31, 44) | -15.152 (1.219) | -13.793 (1.034)

29. Secondary Outcome: Change From Baseline in Blood Biomarker Fibrinogen (Initial Approach)
Description: Biomarker Plasma fibrinogen was determined using the method described by Clauss. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: umol/L
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 35 | 42
umol/L
  Change at Day 7 (n=34, 39) | -3.916 (0.286) | -3.976 (0.261)
  Change at Day 14 (n=33, 38) | 0.404 (0.625) | -0.184 (0.571)
  Change at Day 28 (n=27, 36) | 0.210 (0.676) | 0.014 (0.567)
  Change at Day 56 (n=26, 38) | -2.127 (0.625) | -1.144 (0.515)

30. Secondary Outcome: Change From Baseline in Blood Biomarker Fibrinogen (Extended Approach)
Description: as for outcome 29
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: umol/L
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 45 | 46
umol/L
  Change at Day 7 (n=44, 43) | -3.971 (0.246) | -3.839 (0.244)
  Change at Day 14 (n=43, 42) | 0.051 (0.521) | -0.148 (0.519)
  Change at Day 28 (n=32, 40) | 0.147 (0.599) | -0.091 (0.524)
  Change at Day 56 (n=31, 42) | -2.155 (0.533) | -1.162 (0.462)

31. Secondary Outcome: Change From Baseline in Blood Biomarker Glucose (Initial Approach)
Description: Blood was collected and analyzed for serum glucose levels. A negative change from Baseline indicated improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 37 | 43
mmol/L
  Change at Day 7 (n=37, 41) | 1.617 (0.426) | 1.027 (0.397)
  Change at Day 14 (n=33, 41) | 1.000 (0.300) | 0.432 (0.270)
  Change at Day 28 (n=28, 40) | 0.067 (0.156) | -0.020 (0.129)
  Change at Day 56 (n=27, 40) | 0.255 (0.272) | 0.226 (0.230)

32. Secondary Outcome: Change From Baseline in Blood Biomarker Glucose (Extended Approach)
Description: as for outcome 31
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 47 | 47
mmol/L
  Change at Day 7 (n=46, 45) | 1.767 (0.408) | 0.973 (0.408)
  Change at Day 14 (n=42, 45) | 0.942 (0.254) | 0.364 (0.246)
  Change at Day 28 (n=33, 44) | 0.061 (0.139) | -0.008 (0.119)
  Change at Day 56 (n=32, 43) | 0.189 (0.235) | 0.215 (0.210)

33. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) (Initial Approach)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Pulmonary function testing was performed using spirometry. A positive change from Baseline indicates an improvement. A Mixed Model Repeated Measurement (MMRM) was used for analysis with Baseline value, treatment, visit, and treatment by visit interaction as covariates.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 37 | 43
liters
  Change at Day 7 (n=37, 41) | 0.051 (0.031) | 0.010 (0.029)
  Change at Day 14 (n=33, 41) | 0.083 (0.035) | 0.028 (0.031)
  Change at Day 28 (n=28, 40) | 0.095 (0.037) | 0.001 (0.031)
  Change at Day 56 (n=27, 40) | 0.064 (0.039) | 0.010 (0.033)

34. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) (Extended Approach)
Description: as for outcome 33
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 47 | 47
liters
  Change at Day 7 (n=47, 45) | 0.063 (0.027) | 0.012 (0.028)
  Change at Day 14 (n= 43, 45) | 0.062 (0.029) | 0.018 (0.029)
  Change at Day 28 (n=33, 44) | 0.084 (0.031) | -0.003 (0.028)
  Change at Day 56 (n=32, 44) | 0.050 (0.034) | 0.005 (0.030)

35. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) (Initial Approach)
Description: Forced vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Pulmonary function testing was performed using spirometry. A positive change from Baseline indicates an improvement. A Mixed Model Repeated Measurement (MMRM) was used for analysis with Baseline value, treatment, visit, and treatment by visit interaction as covariates.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 37 | 43
liters
  Change at Day 7 (n=37, 41) | 0.002 (0.060) | 0.057 (0.056)
  Change at Day 14 (n=33, 41) | 0.039 (0.062) | 0.166 (0.056)
  Change at Day 28 (n=28, 40) | 0.039 (0.072) | 0.075 (0.062)
  Change at Day 56 (n=27, 40) | 0.044 (0.072) | 0.086 (0.062)

36. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) (Extended Approach)
Description: as for outcome 35
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 47 | 47
liters
  Change at Day 7 (n=47, 45) | 0.048 (0.052) | 0.062 (0.053)
  Change at Day 14 (n=43, 45) | 0.046 (0.054) | 0.146 (0.053)
  Change at Day 28 (n=33, 44) | 0.053 (0.062) | 0.067 (0.057)
  Change at Day 56 (n=32, 44) | 0.034 (0.065) | 0.084 (0.058)

37. Secondary Outcome: Change From Baseline in FEV1/FVC (Initial Approach)
Description: FEV1/FVC is the percentage of the vital capacity which is expired in the first second of maximal expiration. In healthy patients the FEV1/FVC is usually around 70%. A positive change from Baseline indicates an improvement. A Mixed Model Repeated Measurement (MMRM) was used for analysis with Baseline value, treatment, visit, and treatment by visit interaction as covariates.
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 37 | 43
percent
  Change at Day 7 (n=37, 41) | 1.575 (0.933) | -1.064 (0.870)
  Change at Day 14 (n=33, 41) | 1.874 (1.012) | -1.796 (0.914)
  Change at Day 28 (n=28, 40) | 2.350 (1.138) | -1.029 (0.982)
  Change at Day 56 (n=27, 40) | 1.636 (0.951) | -1.669 (0.828)

38. Secondary Outcome: Change From Baseline in FEV1/FVC (Extended Approach)
Description: as for outcome 37
Time Frame: Baseline and Day 7, Day 14, Day 28 and Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 47 | 47
percent
  Change at Day 7 (n=47, 45) | 1.282 (0.795) | -1.128 (0.799)
  Change at Day 14 (n=43, 45) | 1.394 (0.850) | -1.830 (0.834)
  Change at Day 28 (n=33, 44) | 2.045 (0.974) | -1.198 (0.888)
  Change at Day 56 (n=32, 44) | 1.393 (0.827) | -1.881 (0.765)

39. Secondary Outcome: Chronic Obstructive Pulmonary Assessment Test (CAT) Weekly Averages (Initial Approach)
Description: The CAT is a short, validated, patient-completed questionnaire to assess the impact of COPD on health status. It comprises 8 questions that cover a broad range of effects of COPD on patients' health. Each question is scored in a range between 0 and 5, with the higher end indicating a higher impact of COPD on the patient's wellbeing. The CAT Total score ranges from 0 best) to 40 (Worst).
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
score on a scale
  Week 1 (n=27, 34) | 19.4 (6.65) | 19.2 (7.20)
  Week 2 (n=28, 36) | 17.1 (7.86) | 17.1 (7.48)
  Week 3 (n=24, 37) | 15.9 (7.84) | 16.0 (7.90)
  Week 4 (n=23, 38) | 15.1 (7.85) | 15.8 (8.42)
  Week 5 (n=21, 37) | 14.2 (7.41) | 14.9 (8.04)
  Week 6 (n=19, 37) | 12.9 (6.85) | 15.4 (8.23)
  Week 7 (n=20, 33) | 13.9 (8.93) | 14.7 (8.48)
  Week 8 (n=18, 30) | 12.8 (7.85) | 15.6 (8.25)

40. Secondary Outcome: Chronic Obstructive Pulmonary Assessment Test (CAT) Weekly Averages (Extended Approach)
Description: as for outcome 39
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
score on a scale
  Week 1 (n=37, 38) | 20.4 (7.26) | 19.3 (7.03)
  Week 2 (n=37, 40) | 18.2 (8.54) | 17.2 (7.32)
  Week 3 (n=29, 41) | 16.2 (8.08) | 16.1 (7.73)
  Week 4 (n=27, 42) | 16.0 (8.21) | 15.9 (8.26)
  Week 5 (n=25, 41) | 14.0 (7.28) | 15.1 (7.93)
  Week 6 (n=23, 41) | 12.9 (6.58) | 15.4 (8.12)
  Week 7 (n=24, 37) | 13.5 (8.38) | 14.8 (8.44)
  Week 8 (n=19, 30) | 13.0 (7.68) | 15.6 (8.25)

41. Secondary Outcome: Change From Stable State in Chronic Obstructive Pulmonary Assessment Test (CAT) Weekly Averages (Initial Approach)
Description: The CAT is a short, validated, patient-completed questionnaire to assess the impact of COPD on health status. It comprises 8 questions that cover a broad range of effects of COPD on patients' health. Each question is scored in a range between 0 and 5, with the higher end indicating a higher impact of COPD on the patient's wellbeing. The CAT Total score ranges from 0 best) to 40 (Worst). A negative change from Baseline indicates improvement. Covariates for MMRM are stable state value, treatment, time point, and treatment by time point interaction.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
score on a scale
  Change at Week 1 (n=27, 34) | 6.448 (1.503) | 2.695 (1.096)
  Change at Week 2 (n=28, 36) | 3.778 (1.239) | 0.804 (0.911)
  Change at Week 3 (n=24, 37) | 2.002 (0.915) | 0.278 (0.669)
  Change at Week 4 (n=23, 38) | 0.559 (0.739) | 0.277 (0.536)
  Change at Week 5 (n=21, 37) | -0.412 (0.613) | -0.392 (0.448)
  Change at Week 6 (n=19, 37) | -0.924 (0.411) | -0.062 (0.297)
  Change at Week 7 (n=20, 33) | -0.228 (0.342) | 0.048 (0.253)
  Change at Week 8 (n=18, 30) | 0.002 (0.059) | -0.048 (0.044)

42. Secondary Outcome: Change From Stable State in Chronic Obstructive Pulmonary Assessment Test (CAT) Weekly Averages (Extended Approach)
Description: as for outcome 41
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
scores on a scale
  Week 1 (n=37, 38) | 6.232 (1.424) | 3.009 (1.052)
  Week 2 (n=37, 40) | 3.558 (1.178) | 1.074 (0.876)
  Week 3 (n=29, 41) | 2.044 (0.847) | 0.458 (0.627)
  Week 4 (n=27, 42) | 0.545 (0.732) | 0.429 (0.534)
  Week 5 (n=25, 41) | -0.347 (0.621) | -0.170 (0.459)
  Week 6 (n=23, 41) | -0.668 (0.402) | -0.043 (0.295)
  Week 7 (n=24, 37) | -0.121 (0.310) | 0.014 (0.232)
  Week 8 (n=19, 30) | -0.010 (0.061) | -0.031 (0.045)

43. Secondary Outcome: Exacerbations of Chronic Pulmonary Disease Test (EXACT-PRO) Weekly Averages (Initial Approach)
Description: The EXACT-PRO questionnaire is a new, validated, and standardized measure to evaluate the frequency, severity, and duration of COPD exacerbations. It is a 14-item daily diary, and scores range from 0 to 100, with higher scores indicating worse health status.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
score on a scale
  Week 1 (n=25, 35) | 45.2 (8.54) | 45.1 (8.50)
  Week 2 (n=28, 36) | 41.2 (11.39) | 42.4 (9.07)
  Week 3 (n=24, 38) | 38.8 (11.22) | 40.0 (10.22)
  Week 4 (n=23, 38) | 38.3 (11.00) | 40.2 (11.26)
  Week 5 (n=21, 37) | 35.9 (11.11) | 39.1 (10.55)
  Week 6 (n=19, 37) | 35.1 (9.75) | 39.4 (11.05)
  Week 7 (n=20, 34) | 35.6 (13.69) | 38.7 (12.05)
  Week 8 (n=18, 32) | 34.4 (11.50) | 39.4 (11.34)

44. Secondary Outcome: Exacerbations of Chronic Pulmonary Disease Test (EXACT-PRO) Weekly Averages (Extended Approach)
Description: as for outcome 43
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
score on a scale
  Week 1 (n=35, 39) | 45.6 (9.19) | 45.0 (8.39)
  Week 2 (n=37, 40) | 42.0 (11.07) | 42.3 (8.81)
  Week 3 (n=29, 42) | 39.0 (11.27) | 39.9 (9.82)
  Week 4 (n=27, 42) | 38.8 (11.37) | 40.3 (10.90)
  Week 5 (n=25, 41) | 35.3 (11.03) | 39.1 (10.13)
  Week 6 (n=23, 41) | 33.9 (10.45) | 39.4 (10.62)
  Week 7 (n=24, 38) | 34.3 (13.09) | 38.7 (11.52)
  Week 8 (n=19, 33) | 34.0 (11.30) | 39.6 (11.25)

45. Secondary Outcome: Change From Stable State in Exacerbations of Chronic Pulmonary Disease Test (EXACT-PRO) Weekly Averages (Initial Approach)
Description: The EXACT-PRO questionnaire is a new, validated, and standardized measure to evaluate the frequency, severity, and duration of COPD exacerbations. It is a 14-item daily diary, and scores range from 0 to 100, with higher scores indicating worse health status. A negative change from Baseline indicates improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are baseline value, treatment, time point, treatment by time point and baseline by time point interaction.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
score on a scale
  Change at Week 1 (n=25, 35) | 6.182 (3.271) | 4.753 (2.385)
  Change at Week 2 (n=28, 36) | 4.423 (2.538) | 1.558 (1.864)
  Change at Week 3 (n=24, 38) | 2.080 (2.041) | 0.317 (1.494)
  Change at Week 4 (n=23, 38) | 0.002 (2.003) | 0.657 (1.459)
  Change at Week 5 (n=21, 37) | -1.058 (1.748) | -0.307 (1.276)
  Change at Week 6 (n=19, 37) | -1.688 (1.015) | -0.002 (0.738)
  Change at Week 7 (n=20, 34) | -0.773 (0.698) | 0.002 (0.514)
  Change at Week 8 (n=18, 32) | -0.190 (0.259) | -0.154 (0.191)

46. Secondary Outcome: Change From Stable State in Exacerbations of Chronic Pulmonary Disease Test (EXACT-PRO) Weekly Averages (Extended Approach)
Description: as for outcome 45
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
scores on a scale
  Week 1 (n=35, 39) | 7.163 (2.859) | 4.697 (2.077)
  Week 2 (n=37, 40) | 4.839 (2.259) | 1.433 (1.652)
  Week 3 (n=29, 42) | 2.988 (1.870) | 0.179 (1.363)
  Week 4 (n=27, 42) | 0.909 (1.861) | 0.743 (1.344)
  Week 5 (n=25, 41) | -0.657 (1.554) | -0.318 (1.129)
  Week 6 (n=23, 41) | -0.889 (0.976) | -0.140 (0.706)
  Week 7 (n=24, 38) | -0.311 (0.654) | -0.075 (0.479)
  Week 8 9n=19, 33) | -0.240 (0.244) | -0.115 (0.178)

47. Secondary Outcome: Change From Stable State in Diaries Peak Expiratory Flow (PEF) Weekly Average (Initial Approach)
Description: Morning post-medication PEF (the best of 3 attempts measured with a mini-Wright peak-flow meter) was recorded in a daily diary. A positive change from Baseline indicates improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are stable state value, treatment, time point, and treatment by time point interaction.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
liters/minute
  Change at Week 1 (n=37, 38) | -16.551 (5.144) | -9.915 (4.442)
  Change at Week 2 (n=35, 40) | -6.067 (4.564) | -0.304 (3.899)
  Change at Week 3 (n=35, 40) | -4.996 (3.914) | 0.687 (3.360)
  Change at Week 4 (n=29, 39) | -4.595 (3.421) | -0.420 (2.737)
  Change at Week 5 (n=28, 38) | -3.557 (4.061) | -1.224 (3.287)
  Change at Week 6 (n=27, 37) | -3.795 (4.546) | -5.559 (3.680)
  Change at Week 7 (n=27, 36) | -7.178 (5.212) | -4.186 (4.264)
  Change at Week 8 (n=27, 35) | -2.877 (5.388) | -0.956 (4.418)

48. Secondary Outcome: Change From Stable State in Diaries Peak Expiratory Flow (PEF) Weekly Average (Extended Approach)
Description: as for outcome 47
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
liters/minute
  Change at Week 1 (n=46, 42) | -13.958 (4.147) | -8.447 (3.865)
  Change at Week 2 (n=44, 44) | -5.776 (3.772) | 1.029 (3.488)
  Change at Week 3 (n=44, 44) | -5.360 (3.676) | 2.038 (3.421)
  Change at Week 4 (n=37, 43) | -6.660 (3.546) | 1.133 (3.126)
  Change at Week 5 (n=33, 42) | -5.568 (3.847) | 0.269 (3.396)
  Change at Week 6 (n=32, 41) | -2.186 (3.515) | -4.596 (3.076)
  Change at Week 7 (n=31, 40) | -8.513 (4.544) | -1.974 (3.952)
  Change at Week 8 (n=31, 39) | -4.563 (4.741) | 0.950 (4.091)

49. Secondary Outcome: Change From Stable State in Diaries Symptom Score Weekly Average (Initial Approach)
Description: Any increase in the following respiratory symptoms: dyspnea, sputum purulence, sputum amount, wheeze, sore throat, cough, fever, symptoms of a common cold, ie, nasal congestion and discharge over the previous 24 hours were recorded in a daily diary. Diaries Symptom Score range from 0 to 100, with higher scores indicating worse health status. A negative change from Baseline indicates improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are stable state value, treatment, time point, and treatment by time point interaction.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
score on a scale
  Change at Week 1 (n=38, 42) | 2.930 (0.286) | 2.587 (0.254)
  Change at Week 2 (n=37, 42) | 1.130 (0.314) | 1.331 (0.272)
  Change at Week 3 (n=35, 42) | 0.906 (0.299) | 0.790 (0.258)
  Change at Week 4 (n=30, 40) | 0.552 (0.298) | 0.922 (0.248)
  Change at Week 5 (n=29, 39) | 0.413 (0.305) | 0.882 (0.254)
  Change at Week 6 (n=28, 39) | 0.141 (0.310) | 0.681 (0.258)
  Change at Week 7 (n=27, 37) | 0.442 (0.294) | 0.673 (0.243)
  Change at Week 8 (n=27, 36) | 0.626 (0.361) | 0.612 (0.297)

50. Secondary Outcome: Change From Stable State in Diaries Symptom Score Weekly Average (Extended Approach)
Description: as for outcome 49
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
score on a scale
  Change at Week 1 (n=48, 46) | 3.110 (0.257) | 2.593 (0.246)
  Change at Week 2 (n=47, 46) | 1.171 (0.285) | 1.402 (0.267)
  Change at Week 3 (n=44, 46) | 0.850 (0.267) | 0.802 (0.250)
  Change at Week 4 (n=38, 44) | 0.751 (0.312) | 0.924 (0.282)
  Change at Week 5 (n=34, 43) | 0.437 (0.287) | 0.907 (0.259)
  Change at Week 6 (n=33, 43) | 0.041 (0.257) | 0.661 (0.231)
  Change at Week 7 (n=31, 41) | 0.503 (0.247) | 0.533 (0.216)
  Change at Week 8 (n=31, 40) | 0.451 (0.274) | 0.530 (0.237)

51. Secondary Outcome: Change From Stable State in Diaries Treatment Score Weekly Average (Initial Approach)
Description: Any changes in the participant's usual treatment were recorded in a daily diary. Diaries Symptom Score range from 0 to 100, with higher scores indicating worse health status. A negative change from Baseline indicates improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are stable state value, treatment, time point, and treatment by time point interaction.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
score on a scale
  Change at Week 1 (n=38, 42) | 0.849 (0.194) | 0.769 (0.174)
  Change at Week 2 (n=37, 42) | 0.682 (0.190) | 0.804 (0.167)
  Change at Week 3 (n=35, 42) | 0.281 (0.115) | 0.188 (0.099)
  Change at Week 4 (n=30, 40) | 0.185 (0.118) | 0.217 (0.099)
  Change at Week 5 (n=29, 39) | 0.130 (0.123) | 0.263 (0.103)
  Change at Week 6 (n=28, 39) | 0.128 (0.130) | 0.204 (0.108)
  Change at Week 7 (n=27, 37) | 0.112 (0.117) | 0.135 (0.097)
  Change at Week 8 (n=27, 36) | 0.122 (0.101) | 0.127 (0.084)

52. Secondary Outcome: Change From Stable State in Diaries Treatment Score Weekly Average (Extended Approach)
Description: as for outcome 51
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
score on a scale
  Change at Week 1 (n=48, 46) | 0.787 (0.170) | 0.730 (0.162)
  Change at Week 2 (n=47, 46) | 0.767 (0.172) | 0.780 (0.161)
  Change at Week 3 (n=44, 46) | 0.338 (0.103) | 0.177 (0.095)
  Change at Week 4 (n=38, 44) | 0.379 (0.144) | 0.206 (0.129)
  Change at Week 5 (n=34, 43) | 0.191 (0.107) | 0.244 (0.096)
  Change at Week 6 (n=33, 43) | 0.127 (0.107) | 0.196 (0.096)
  Change at Week 7 (n=31, 41) | 0.179 (0.116) | 0.156 (0.103)
  Change at Week 8 (n=31, 40) | 0.084 (0.086) | 0.171 (0.075)

53. Secondary Outcome: Change From Stable State in Diaries Hours Out of the Home Weekly Average (Initial Approach)
Description: Estimates of the length of time the participants were out of their own home on the previous day were recorded in a daily diary. A negative change from Baseline indicates improvement. Covariates for Mixed Model Repeated Measurement (MMRM) are stable state value, treatment, time point, and treatment by time point interaction.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
hours
  Change at Week 1 (n=34, 34) | -1.313 (0.416) | -0.105 (0.391)
  Change at Week 2 (n=34, 38) | -0.974 (0.359) | -0.328 (0.333)
  Change at Week 3 (n=34, 40) | -1.077 (0.374) | 0.226 (0.335)
  Change at Week 4 (n=28, 39) | -1.131 (0.414) | -0.306 (0.354)
  Change at Week 5 (n=26, 38) | -0.826 (0.465) | 0.280 (0.407)
  Change at Week 6 (n=25, 35) | -1.154 (0.448) | -0.062 (0.386)
  Change at Week 7 (n=26, 35) | -1.194 (0.449) | -0.340 (0.394)
  Change at Week 8 (n=26, 34) | -0.812 (0.532) | 0.037 (0.458)

54. Secondary Outcome: Change From Stable State in Diaries Hours Out of the Home Weekly Average (Extended Approach)
Description: as for outcome 53
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7 and 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
hours
  Change at Week 1 (n=42, 38) | -1.472 (0.353) | -0.276 (0.344)
  Change at Week 2 (n=43, 42) | -1.305 (0.319) | -0.472 (0.307)
  Change at Week 3 (n=42, 44) | -1.314 (0.343) | 0.099 (0.324)
  Change at Week 4 (n=35, 43) | -1.328 (0.357) | -0.266 (0.325)
  Change at Week 5 (n=31, 42) | -0.833 (0.402) | 0.158 (0.369)
  Change at Week 6 (n=30, 39) | -1.271 (0.372) | -0.247 (0.344)
  Change at Week 7 (n=30, 39) | -1.144 (0.363) | -0.478 (0.333)
  Change at Week 8 (n=30, 38) | -0.714 (0.443) | -0.068 (0.401)

55. Secondary Outcome: Exacerbation Length (Initial Approach)
Description: Exacerbation length is the period from start of increased symptoms to end of increased symptoms; the last day of an exacerbation was to be followed by 2 days without symptom entries in the diary.
Time Frame: 8 Weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 38 | 43
days | 12.0 [8.0 to 18.0] | 14.0 [10.0 to 17.0]

56. Secondary Outcome: Exacerbation Length (Extended Approach)
Description: as for outcome 55
Time Frame: 8 Weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 48 | 47
days | 13.0 [9.0 to 19.0] | 14.0 [11.0 to 17.0]

57. Secondary Outcome: Change From Baseline in Aortic Pulse Wave Velocity in a Subset of Participants (Initial Approach)
Description: Carotid-femoral aortic pulse wave velocity (aPWV) will be measured in a subset of participants to determine changes in arterial stiffness. A negative change from Baseline indicates improvement. Covariates for MMRM are baseline value, treatment, visit, and treatment by visit interaction.
Time Frame: Baseline and Days 14 and 28
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: meters/second
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 24 | 28
meters/second
  Change at Day 14 (n=18, 24) | -0.047 (0.337) | -0.343 (0.290)
  Change at Day 28 (n=14, 24) | -0.380 (0.413) | -0.474 (0.321)

58. Secondary Outcome: Change From Baseline in Aortic Pulse Wave Velocity in a Subset of Participants (Extended Approach)
Description: as for outcome 57
Time Frame: Baseline and Days 14 and 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: meters/second
Arm/Group | Roflumilast 500 μg | Placebo
Number analyzed (Participants) | 34 | 32
meters/second
  Change at Day 14 (n=28, 28) | -0.128 (0.247) | -0.326 (0.245)
  Change at Day 28 (n=19, 28) | -0.316 (0.323) | -0.511 (0.273)

ADVERSE EVENTS:
Time Frame: Signing of informed consent until Follow-up Visit (Up to 56 days)
Description: AEs were analyzed using an Initial Approach (all patients treated in Cycle 1) and an Extended Approach (all patients treated in Cycle 1 and patients re-randomized and treated in Cycle 2). The data from the 2 approaches are entered in one table. Please note: a result of 0 corresponds to no patients with AEs for the preferred term > the 5% threshold.
Groups:
- Roflumilast 500 μg (Initial Approach): Roflumilast 500 µg tablet, once daily, orally in the morning after breakfast added on to standard therapy for acute COPD exacerbations. Initial Approach Arm includes all participants who received treatment in Cycle 1.
- Placebo (Initial Approach): Placebo matching roflumilast tablet, once daily, orally in the morning after breakfast added on to standard therapy for acute COPD exacerbations. Initial Approach Arm includes all participants who received treatment in Cycle 1.
- Roflumilast 500 µg (Extended Approach): Roflumilast 500 µg tablet, once daily, orally in the morning after breakfast added on to standard therapy for acute COPD exacerbations. Extended Approach Arm includes all participants who received treatment in Cycle 1 and those participants who were re-randomized and received treatment in Cycle 2.
- Placebo (Extended Approach): Placebo matching roflumilast tablet, once daily, orally in the morning after breakfast added on to standard therapy for acute COPD exacerbations. Extended Approach Arm includes all participants who received treatment in Cycle 1 and those participants who were re-randomized and received treatment in Cycle 2.
Arm/Group | Roflumilast 500 μg (Initial Approach) | Placebo (Initial Approach) | Roflumilast 500 µg (Extended Approach) | Placebo (Extended Approach)
Serious Adverse Events (participants affected / at risk) | 4/38 | 1/43 | 4/48 | 1/47
Other Adverse Events (participants affected / at risk) | 35/38 | 25/43 | 44/48 | 28/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast 500 μg (Initial Approach) (N=38) | Placebo (Initial Approach) (N=43) | Roflumilast 500 µg (Extended Approach) (N=48) | Placebo (Extended Approach) (N=47)
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast 500 μg (Initial Approach) (N=38) | Placebo (Initial Approach) (N=43) | Roflumilast 500 µg (Extended Approach) (N=48) | Placebo (Extended Approach) (N=47)
Diarrhoea (Gastrointestinal disorders) | 25 | 10 | 32 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 6 | 3 | 9 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 6 | 2
Dizziness (Nervous system disorders) | 6 | 1 | 6 | 1
Headache (Nervous system disorders) | 3 | 2 | 4 | 2
Insomnia (Psychiatric disorders) | 12 | 2 | 14 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 | 13 | 19 | 15
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.